CLINICAL TRIAL: NCT06605859
Title: An Open, Multicentre, Prospective, Non-interventional Study of the CE-marked Medical Device GlucoTab in Nursing Homes and Domiciliary Nursing Care, According to Intended Use Without Additional Invasive and Stressful Measures
Brief Title: DigiDiab Pilot Spain - Nursing Home and Domiciliary Nursing Care
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 230206 EIT Health-nursing home
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
Keywords: GlucoTab; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GlucoTab Prospective Group
  Interventions: Device: GlucoTab
- Retrospective Control Group
  Interventions: Other: Diabetes Treatment

INTERVENTIONS:
Device: GlucoTab — Insulin therapy will be started and adjusted according to the GlucoTab system with incorporated software algorithm. The goal of the basal-insulin algorithm is to maintain blood glucose within acceptable targets according to the predefined health status.
  For a limited time period after therapy start, three measurements per day are suggested by the algorithm to determine blood glucose. Insulin dosage titration will be performed according to the algorithm in GlucoTab under supervision of the nurses of the nursing homes/domiciliary nursing care. Correctional bolus insulin will be administered at defined time-points according to BG targets in the predefined health status.
  Nurses and nursing assistants will be trained in the use of the GlucoTab.
  Groups: GlucoTab Prospective Group
Other: Diabetes Treatment — Diabetes Standard Care
  Groups: Retrospective Control Group

SUMMARY:
GlucoTab is a stand-alone software system to support healthcare professionals in the care of patients with diabetes mellitus or newly diagnosed hyperglycaemia who are treated with insulin and/or other glucose-lowering drugs or of patients only requiring glucose monitoring.

It provides a therapy algorithm for subcutaneous basal insulin therapy of patients with type 2 diabetes, which will be used in this study.

DETAILED DESCRIPTION:
GlucoTab: The CE-marked medical device GlucoTab is a system designed to support healthcare personnel in managing insulin therapy for patients with diabetes.

In this study, only the GlucoTab algorithm supported basalinsulin therapy will be used, which is intended for patients with Type 2 diabetes in domiciliary nursing care and nursing homes requiring insulin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Elderly people, willing to be treated with a basal insulin therapy according to the GlucoTab system
* Informed consent obtained after being advised of the nature of the study
* Male or female aged ≥ 18 years
* Type 2 diabetes (treated with insulin therapy)
* Residents of participating nursing homes/domiciliary nursing care in the region of Camp de Tarragona (Spain).

Exclusion Criteria:

* type 1 diabetes mellitus
* intravenous insulin therapy
* hyperglycaemic episodes (ketoacidosis, hyperosmolar state) if they require intravenous insulin therapy
* continuous subcutaneous insulin infusion
* gestational diabetes or pregnancy
* known or suspected allergy to insulin
* total parenteral nutrition
* any mental condition rendering the patient incapable of giving his/her consent
* any disease or condition which according to the investigator would interfere with the trial or the safety of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-critically ill patients with type 2 diabetes in the participating nursing homes/domiciliary nursing care who require s.c. insulin therapy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Efficacy - mean percentage of fasting blood glucose in target range | ≥ 24 hours after start of the therapy by using the GlucoTab system
  Efficacy is assessed by evaluating the Mean percentage of Fasting Blood Glucose in the target range 80 - 180 mg/dl

SECONDARY OUTCOMES:
Usability | at the end of the study, on average three months
  adherence to dose suggestions of the GlucoTab system
Safety - number of hypoglycaemic events | at the end of the study, on average three months
  Safety is assessed by evaluating the number of hypoglycaemic events
Efficacy - mean pre-breakfast blood glucose | at the end of the study, on average three months
  mean pre-breakfast blood glucose

CONTACTS AND LOCATIONS:
Locations (1):
- IDIAP Jordi Gol, Tarragona, Spain